CLINICAL TRIAL: NCT00784979
Title: Reduction of PRA (Panel Reactive Antibody) in Sensitized Patients Awaiting Live-Donor Renal Transplantation
Brief Title: Panel Reactive Antibody (PRA) Reduction in Sensitized Patients Awaiting Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampa General Hospital (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS_100109
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: End Stage Renal Disease
Keywords: Renal; Transplant; PRA
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — cytomegalovirus-specific hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CMVIG followed by PP (No Intervention): MMF or rapamycin was given with CMVIG for 4 weeks followed by plasmapheresis
  Interventions: Drug: CMVIG

INTERVENTIONS:
Drug: CMVIG — 400mg/kg IV (60mg/kg/IV/hr initially, titrated up) once a week up to four weeks
  Other Names: Cytomegalovirus Immune Globulin - Intravenous; Cytogam

SUMMARY:
The purpose of this study is to offer Panel Reactive Antibodies [PRA] reduction treatment to high responder renal transplant patients who otherwise may never be compatible with a potential organ donor. PRA reduction is offered in the following phases:

1. Immunological Testing
2. Transplant Nephrectomy
3. Pharmacologic Therapy
4. Plasmapheresis
5. Transplant

DETAILED DESCRIPTION:
Patients with high level of preformed antibodies (panel reactive antibodies [PRA]) to donor antigens make identification of a suitable donor difficult. For most transplant centers, 20-35% of patients waiting for a kidney transplant comprise this challenging group. These patients have a wait time of over five years and have many incompatible cross-matches with potential organ donors.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients with a potential living donor who is incompatible (T-&/or B-cell locus) due to recipient high PRA or MHC antibodies
* PRA greater than or equal to 20% within last twelve months
* Recipient and donor accepted as potential candidates by the LifeLink Healthcare Renal Transplant Committee

Exclusion Criteria:

* Patients with known allergy to CytoGam(R), Cellcept, Rapamycin
* Patients who will receive IVIG or CytoGam(R) for any cause prior to protocol process
* ABO incompatibility
* Patients not capable of following through the treatment for various reasons as determined by treating physicians
* Any potential recipient who is pregnant or becomes pregnant
* Exclusion for Plasmapheresis: known allergy to ethylene oxide or natural rubber latex.
* Exclusion for Plasmapheresis: Intake of ACE-inhibitor or Angtiotensiin-receptor blockers in the last 24 hours prior to plasma exchange

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-01; Primary Completion 2010-12 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Leone, MD, PhD, Principal Investigator — Lifelink Healthcare Institute
Locations (1):
- LifeLink HealthCare Institute, Tampa, Florida, United States

REFERENCES:
- See also: Tampa General Medical Group — http://www.tgmg.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CMVIG Followed by PP
Started | 26
Completed | 20
Not Completed | 6
Not completed — incomplete data | 6

BASELINE CHARACTERISTICS:
Groups:
- Highly Sensitized Patients: Highly-sensitized patients were defined as those having PRA >/= 20% within the last 12 months; identification of donor-specific antibody or, any combination of Class I and/or Class 2 HLA incompatibility.
Arm/Group | Highly Sensitized Patients
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — >/= 18 years old
  years | 42 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Percent of subjects with PRA >/= 20% in last 12 months [Number; unit: percent of subjects with elevated PRA] | 76

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Sensitized Patients Treated With PRA Reduction Pharmacological Therapy, Including Cytogam, Who Become Cross-match Compatible With Potential Living Donor
Description: The percent of sensitized patients treated with PRA Reduction Pharmacological Therapy, including Cytogam, who become cross-match compatible with potential living donor. Treatment success defined as achieving a decrease in donor specific antibody and eliminating cross-match incompatibility sufficient to allow transplantation.
Time Frame: four weeks
Measure: Number; unit: percent of subjects becoming compatible
Groups:
- Highly Sensitized Patients: Highly-sensitized patients were defined as those having PRA greater than or equal to 20 percent within the last 12 months, identification of donor-specific antibody or, any combination of Class I and/or Class 2 HLA incompatibility.
Arm/Group | Highly Sensitized Patients
Number analyzed (Participants) | 20
percent of subjects becoming compatible | 40

2. Secondary Outcome: Monitor Graft Survival
Time Frame: 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Monitor Patient Survival
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Highly Sensitized Patients
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes